CLINICAL TRIAL: NCT03147274
Title: Evaluation of a Group Curriculum to Improve Self-Management Adherence and Transition Readiness in Older Teens With Type 1 Diabetes
Brief Title: Group Education Curriculum for Older Teens With Type 1 Diabetes
Acronym: SMART T1D
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Katharine Garvey, Pediatric Endocrinologist, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB-P00023671
Record Dates: First submitted 2017-05-05; First posted 2017-05-10 (Actual); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Diabetes Mellitus, Type 1; Adolescence
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Methods

STUDY DESIGN:
Intervention Model Description: This is a 12-month randomized controlled trial evaluating the impact of a health care delivery intervention ("SMART T1D" - a 3-session group educational curriculum), compared to standard care, on self-care adherence and transition readiness in adolescents with type 1 diabetes. Intervention (group sessions) and control (standard care) subjects will complete the study on a parallel timeline.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Participants in this group will receive 3 group education sessions led by a diabetes nurse educator in addition to standard care.
  Interventions: Behavioral: Intervention
- Control Group (No Intervention): These participants will receive no intervention. They will have clinic care as usual and will receive three diabetes newsletters to match for attention.

INTERVENTIONS:
Behavioral: Intervention — Patients randomized to the intervention group will attend 3 SMART T1D group curriculum sessions over the study period, in addition to usual diabetes clinic care. Each interactive group session will last 2 hours and will be facilitated by a diabetes nurse educator.
  Arms: Intervention Group

SUMMARY:
SMART T1D is a research study that offers interactive diabetes education for teens with type 1 diabetes in peer groups led by diabetes nurse educators. Participants in the study will be randomly assigned to either receive three of the group sessions in addition to their routine clinic care or to receive their usual diabetes clinic care.

DETAILED DESCRIPTION:
The objective of this 12-month pilot randomized controlled trial is to evaluate the impact of a 3-session group educational curriculum, compared to standard care, on self-care adherence and transition readiness in adolescents with type 1 diabetes in the Boston Children's Hospital (BCH) Diabetes Program. Adolescents (15-18 years) with T1D will be randomized to receive a 3-session group curriculum ("SMART T1D" - Self-Management, Adherence and Readiness for Transition in T1D) in addition to usual care (intervention group) or to receive usual care with individual diabetes visits (control group) and electronic newsletters to match for attention.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in the pediatric diabetes clinic at Boston Children's Hospital
* Age 15-18 years at enrollment
* Diabetes duration >1 year
* Ability to speak/read English
* Visits to any BCH Diabetes Program site ≥1 times over the past 6 months
* Hemoglobin A1c at clinic visit prior to enrollment 7.5%-11%

Exclusion Criteria:

* Major medical or psychiatric comorbidities
* Established patients of one of the diabetes nurse educators delivering the intervention

Ages: 15 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2017-05-03 (Actual); Primary Completion 2019-02-21 (Actual); Study Completion 2019-02-21 (Actual)

PRIMARY OUTCOMES:
Change from baseline self-care adherence at 12 months | 12 months
  Measured by the Self-Care Inventory-Revised (SCI-R)

SECONDARY OUTCOMES:
Change from baseline transition readiness at 12 months | 12 months
  Measured by the Readiness for Independent Self-Care Questionnaire (RISQ)
Change from baseline hemoglobin A1c at 12 months | 12 months
  Measured by DCA Vantage

CONTACTS AND LOCATIONS:
Overall Officials: Katharine Garvey, MD, MPH, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared with other researchers

REFERENCES:
- [Background] Bryden KS, Dunger DB, Mayou RA, Peveler RC, Neil HA. Poor prognosis of young adults with type 1 diabetes: a longitudinal study. Diabetes Care. 2003 Apr;26(4):1052-7. doi: 10.2337/diacare.26.4.1052. PMID 12663572
- [Background] Laing SP, Swerdlow AJ, Slater SD, Botha JL, Burden AC, Waugh NR, Smith AW, Hill RD, Bingley PJ, Patterson CC, Qiao Z, Keen H. The British Diabetic Association Cohort Study, I: all-cause mortality in patients with insulin-treated diabetes mellitus. Diabet Med. 1999 Jun;16(6):459-65. doi: 10.1046/j.1464-5491.1999.00075.x. PMID 10391392
- [Background] Jacobson AM, Hauser ST, Willett J, Wolfsdorf JI, Herman L. Consequences of irregular versus continuous medical follow-up in children and adolescents with insulin-dependent diabetes mellitus. J Pediatr. 1997 Nov;131(5):727-33. doi: 10.1016/s0022-3476(97)70101-x. PMID 9403654
- [Background] Wills CJ, Scott A, Swift PG, Davies MJ, Mackie AD, Mansell P. Retrospective review of care and outcomes in young adults with type 1 diabetes. BMJ. 2003 Aug 2;327(7409):260-1. doi: 10.1136/bmj.327.7409.260. No abstract available. PMID 12896937
- [Background] Bryden KS, Peveler RC, Stein A, Neil A, Mayou RA, Dunger DB. Clinical and psychological course of diabetes from adolescence to young adulthood: a longitudinal cohort study. Diabetes Care. 2001 Sep;24(9):1536-40. doi: 10.2337/diacare.24.9.1536. PMID 11522695
- [Background] Laing SP, Jones ME, Swerdlow AJ, Burden AC, Gatling W. Psychosocial and socioeconomic risk factors for premature death in young people with type 1 diabetes. Diabetes Care. 2005 Jul;28(7):1618-23. doi: 10.2337/diacare.28.7.1618. PMID 15983310
- [Background] Lotstein DS, Seid M, Klingensmith G, Case D, Lawrence JM, Pihoker C, Dabelea D, Mayer-Davis EJ, Gilliam LK, Corathers S, Imperatore G, Dolan L, Anderson A, Bell RA, Waitzfelder B; SEARCH for Diabetes in Youth Study Group. Transition from pediatric to adult care for youth diagnosed with type 1 diabetes in adolescence. Pediatrics. 2013 Apr;131(4):e1062-70. doi: 10.1542/peds.2012-1450. Epub 2013 Mar 25. PMID 23530167
- [Background] Helgeson VS, Reynolds KA, Snyder PR, Palladino DK, Becker DJ, Siminerio L, Escobar O. Characterizing the transition from paediatric to adult care among emerging adults with Type 1 diabetes. Diabet Med. 2013 May;30(5):610-5. doi: 10.1111/dme.12067. Epub 2013 Feb 28. PMID 23157171
- [Background] Peters A, Laffel L; American Diabetes Association Transitions Working Group. Diabetes care for emerging adults: recommendations for transition from pediatric to adult diabetes care systems: a position statement of the American Diabetes Association, with representation by the American College of Osteopathic Family Physicians, the American Academy of Pediatrics, the American Association of Clinical Endocrinologists, the American Osteopathic Association, the Centers for Disease Control and Prevention, Children with Diabetes, The Endocrine Society, the International Society for Pediatric and Adolescent Diabetes, Juvenile Diabetes Research Foundation International, the National Diabetes Education Program, and the Pediatric Endocrine Society (formerly Lawson Wilkins Pediatric Endocrine Society). Diabetes Care. 2011 Nov;34(11):2477-85. doi: 10.2337/dc11-1723. No abstract available. PMID 22025785
- [Background] Weissberg-Benchell J, Wolpert H, Anderson BJ. Transitioning from pediatric to adult care: a new approach to the post-adolescent young person with type 1 diabetes. Diabetes Care. 2007 Oct;30(10):2441-6. doi: 10.2337/dc07-1249. Epub 2007 Jul 31. No abstract available. PMID 17666466
- [Background] Holmes-Walker DJ, Llewellyn AC, Farrell K. A transition care programme which improves diabetes control and reduces hospital admission rates in young adults with Type 1 diabetes aged 15-25 years. Diabet Med. 2007 Jul;24(7):764-9. doi: 10.1111/j.1464-5491.2007.02152.x. Epub 2007 May 29. PMID 17535294
- [Background] Van Walleghem N, Macdonald CA, Dean HJ. Evaluation of a systems navigator model for transition from pediatric to adult care for young adults with type 1 diabetes. Diabetes Care. 2008 Aug;31(8):1529-30. doi: 10.2337/dc07-2247. Epub 2008 May 5. PMID 18458141
- [Background] Lane JT, Ferguson A, Hall J, McElligott M, Miller M, Lane PH, Pfeffer E. Glycemic control over 3 years in a young adult clinic for patients with type 1 diabetes. Diabetes Res Clin Pract. 2007 Dec;78(3):385-91. doi: 10.1016/j.diabres.2007.04.014. Epub 2007 Jun 28. PMID 17602780
- [Background] Logan J, Peralta E, Brown K, Moffett M, Advani A, Leech N. Smoothing the transition from paediatric to adult services in type 1 diabetes. J Diabetes Nurs. 2008;12:328-38.
- [Background] Orr DP, Fineberg NS, Gray DL. Glycemic control and transfer of health care among adolescents with insulin dependent diabetes mellitus. J Adolesc Health. 1996 Jan;18(1):44-7. doi: 10.1016/1054-139X(95)00044-S. PMID 8750427
- [Background] American Academy of Pediatrics; American Academy of Family Physicians; American College of Physicians; Transitions Clinical Report Authoring Group; Cooley WC, Sagerman PJ. Supporting the health care transition from adolescence to adulthood in the medical home. Pediatrics. 2011 Jul;128(1):182-200. doi: 10.1542/peds.2011-0969. Epub 2011 Jun 27. PMID 21708806
- [Background] Schwartz LA, Brumley LD, Tuchman LK, Barakat LP, Hobbie WL, Ginsberg JP, Daniel LC, Kazak AE, Bevans K, Deatrick JA. Stakeholder validation of a model of readiness for transition to adult care. JAMA Pediatr. 2013 Oct;167(10):939-46. doi: 10.1001/jamapediatrics.2013.2223. PMID 23959392
- [Background] Schwartz LA, Tuchman LK, Hobbie WL, Ginsberg JP. A social-ecological model of readiness for transition to adult-oriented care for adolescents and young adults with chronic health conditions. Child Care Health Dev. 2011 Nov;37(6):883-95. doi: 10.1111/j.1365-2214.2011.01282.x. PMID 22007989
- [Background] Raymond JK, Berget CL, Driscoll KA, Ketchum K, Cain C, Fred Thomas JF. CoYoT1 Clinic: Innovative Telemedicine Care Model for Young Adults with Type 1 Diabetes. Diabetes Technol Ther. 2016 Jun;18(6):385-90. doi: 10.1089/dia.2015.0425. Epub 2016 May 19. PMID 27196443
- [Background] Raymond JK, Shea JJ, Berget C, Cain C, Fay-Itzkowitz E, Gilmer L, Hoops S, Owen D, Shepard D, Spiegel G, Klingensmith G. A novel approach to adolescents with type 1 diabetes: the team clinic model. Diabetes Spectr. 2015 Jan;28(1):68-71. doi: 10.2337/diaspect.28.1.68. No abstract available. PMID 25717281
- [Background] Floyd BD, Block JM, Buckingham BB, Ly T, Foster N, Wright R, Mueller CL, Hood KK, Shah AC. Stabilization of glycemic control and improved quality of life using a shared medical appointment model in adolescents with type 1 diabetes in suboptimal control. Pediatr Diabetes. 2017 May;18(3):204-212. doi: 10.1111/pedi.12373. Epub 2016 Feb 26. PMID 26919322
- [Background] Lewin AB, LaGreca AM, Geffken GR, Williams LB, Duke DC, Storch EA, Silverstein JH. Validity and reliability of an adolescent and parent rating scale of type 1 diabetes adherence behaviors: the Self-Care Inventory (SCI). J Pediatr Psychol. 2009 Oct;34(9):999-1007. doi: 10.1093/jpepsy/jsp032. Epub 2009 May 7. PMID 19423660
- [Background] Weinger K, Butler HA, Welch GW, La Greca AM. Measuring diabetes self-care: a psychometric analysis of the Self-Care Inventory-Revised with adults. Diabetes Care. 2005 Jun;28(6):1346-52. doi: 10.2337/diacare.28.6.1346. PMID 15920050
- [Background] Sawicki GS, Lukens-Bull K, Yin X, Demars N, Huang IC, Livingood W, Reiss J, Wood D. Measuring the transition readiness of youth with special healthcare needs: validation of the TRAQ--Transition Readiness Assessment Questionnaire. J Pediatr Psychol. 2011 Mar;36(2):160-71. doi: 10.1093/jpepsy/jsp128. Epub 2009 Dec 29. PMID 20040605
- [Background] Welch GW, Jacobson AM, Polonsky WH. The Problem Areas in Diabetes Scale. An evaluation of its clinical utility. Diabetes Care. 1997 May;20(5):760-6. doi: 10.2337/diacare.20.5.760. PMID 9135939
- [Background] Varni JW, Burwinkle TM, Jacobs JR, Gottschalk M, Kaufman F, Jones KL. The PedsQL in type 1 and type 2 diabetes: reliability and validity of the Pediatric Quality of Life Inventory Generic Core Scales and type 1 Diabetes Module. Diabetes Care. 2003 Mar;26(3):631-7. doi: 10.2337/diacare.26.3.631. PMID 12610013
- [Background] Iannotti RJ, Schneider S, Nansel TR, Haynie DL, Plotnick LP, Clark LM, Sobel DO, Simons-Morton B. Self-efficacy, outcome expectations, and diabetes self-management in adolescents with type 1 diabetes. J Dev Behav Pediatr. 2006 Apr;27(2):98-105. doi: 10.1097/00004703-200604000-00003. PMID 16682872
- [Background] Khagram L, Martin CR, Davies MJ, Speight J. Psychometric validation of the Self-Care Inventory-Revised (SCI-R) in UK adults with type 2 diabetes using data from the AT.LANTUS Follow-on study. Health Qual Life Outcomes. 2013 Feb 26;11:24. doi: 10.1186/1477-7525-11-24. PMID 23443007
- [Background] Markowitz JT, Laffel LM. Transitions in care: support group for young adults with Type 1 diabetes. Diabet Med. 2012 Apr;29(4):522-5. doi: 10.1111/j.1464-5491.2011.03537.x. PMID 22150392